CLINICAL TRIAL: NCT03035617
Title: Post-Operative Pain After Laparoscopic Ventral Hernia Repair, Impact of Mesh Impregnation With Bupivacaine Solution vs. Normal Saline Solution
Brief Title: Study to Evaluate Reduction in Pain After Laparoscopic Hernia Repair With Mesh Soaked in Bupivacaine Solution
Acronym: HAPPIEST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Noman Shahzad, Dr, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HAPPIEST Trial
Record Dates: First submitted 2017-01-25; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Abdominal Wall Defect
Keywords: Bupivacaine
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: We propose a parallel design having two arms. In both the arms operative procedure of laparoscopic ventral hernia repair will be the same except solution used to soak the mesh before application. In control arm mesh will be soaked in normal saline solution as is routinely done. In intervention arm mesh will be soaked in .5% bupivacaine solution before application. Twenty ml of .5% bupivacaine will be provided by Institutional Clinical Trial Unit in coded form. Record of the codes will be kept by the clinical trial unit. Soaking will be done for one minute. Participants, investigators and outcome assessors will be blinded of the treatment allocation.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Allocation will be done by the staff at clinical trial unit which will be kept undisclosed to the investigators, patients and outcome assessors. Clinical Trial Unit will provide the solution for soaking mesh in coded form according to treatment arm allocation.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Controlled Arm (Placebo Comparator): Mesh will be soaked in normal saline solution as is routinely done.
  Interventions: Other: Saline
- Intervention Arm (Experimental): Mesh will be soaked in .5% bupivacaine solution before application.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine is long acting local anesthetic drug. Though minimum toxic dose of bupivacaine for intra-peritoneal use is not defined, analgesic effect of its intra-peritoneal use especially after laparoscopic cholecystectomy has been assessed in several interventional studies. Intra-peritoneal use of up to 50ml of .25% , , or up to 20ml of .5% solution has not shown any drug related adverse reactions .
  Arms: Intervention Arm
Other: Saline — In control arm mesh will be soaked in normal saline solution as is routinely done.
  Arms: Controlled Arm

SUMMARY:
Early post-operative pain and discomfort after laparoscopic repair remains a concern for patients requiring hospital stay and parenteral narcotic analgesics . This quite often proves to be a hindrance in early ambulation, enhances patient discomfort and prevents early discharge from hospital.

Local anesthetics infiltration at wound site after various procedures is known to be effective in reducing immediate post-operative pain , . In case of laparoscopic ventral hernia repair, delivering local anesthetic at site of mesh application can be achieved by soaking the mesh in local anesthetic solution before application. To date there is no evidence regarding impact of soaking mesh in bupivacaine solution before application in case of laparoscopic ventral hernia repair.

OBJECTIVE:

Primary Objective:

To evaluate impact of impregnating mesh in .5% bupivacaine solution as compared to normal saline solution on post-operative pain after laparoscopic ventral hernia repair.

Secondary Objective:

To evaluate impact of impregnating mesh in .5% bupivacaine solution as compared to saline solution on length of hospital stay after laparoscopic ventral hernia repair.

Study Sample:

Patients with uncomplicated ventral abdominal wall hernia presenting at general surgery clinics of AKUH Karachi who are planned to undergo laparoscopic repair and meet eligibility criteria of inclusion into trial.

SETTINGS:

Study will be conducted in General Surgery Section of Aga Khan University Hospital, Karachi.

Patients will be evaluated in clinic at the time of presentation regarding eligibility to participate in study. Written informed consent will be taken in clinic. A copy of the consent form will be handed over to the patient. Clinical Trial Unit will be informed of the scheduled date and time of the operation. Allocation will be done by the staff at clinical trial unit which will be kept undisclosed to the investigators, patients and outcome assessors. Clinical Trial Unit will provide the solution for soaking mesh in coded form according to treatment arm allocation. After the operation first assessment of pain will be done six hours post-operatively using VAS. Second assessment will be done at twenty four hours from end of operation. This assessment will be done directly if patient is admitted in the hospital or will be done on telephone if patient is discharged home.

FOLLOW UP:

Pain assessment will be done using visual analogue scale (VAS). This is validated score to measure level of pain. It ranges from zero to ten. Score of 0 means no pain and score of ten means worst pain one can ever have. Score will be assessed at 6 and 24 hours from procedure.

DETAILED DESCRIPTION:
INTRODUCTION:

Laparoscopic approach to uncomplicated ventral hernia repair as compared to open repair has advantages of less post operative pain, less rates of wound infection , , early recovery, shortened hospital stay and less overall cost of treatment , , . Patient satisfaction after laparoscopic procedure is better as compared to open repair . Recurrence rate is also known to be less in laparoscopic repair as compared to open repair. Despite all this, laparoscopic approach is utilized in only about quarter of patients with ventral hernia in developed countries , . Early post-operative pain and discomfort after laparoscopic repair remains a concern for patients requiring hospital stay and parenteral narcotic analgesics . Intensity of pain is similar regardless of method of fixation of mesh. This quite often proves to be a hindrance in early ambulation, enhances patient discomfort and prevents early discharge from hospital. Early post-operative pain is thought to be secondary to dissection in the area of mesh application. Local application of anesthetic agent is this area can potentially overcome this problem and make the procedure feasible as an ambulatory care operation.

Local anesthetics infiltration at wound site after various procedures is known to be effective in reducing immediate post-operative pain , . In case of laparoscopic ventral hernia repair, delivering local anesthetic at site of mesh application can be achieved by soaking the mesh in local anesthetic solution before application. Bupivacaine is long acting local anesthetic. Results of studies that have used this class of drugs intra-peritonealy in other types of surgeries for analgesic purpose have shown it to be safe for intra-operative use. To date there is no evidence regarding impact of soaking mesh in bupivacaine solution before application in case of laparoscopic ventral hernia repair. These patients require post operative intravenous analgesic agents to deal with early post operative pain.

If this turns out to be effective intervention, it will improve patient satisfaction and early discharge from hospital. This can also potentially reduce cost of care.

OBJECTIVE:

Primary Objective:

To evaluate impact of impregnating mesh in .5% bupivacaine solution as compared to normal saline solution on post-operative pain after laparoscopic ventral hernia repair.

Secondary Objective:

To evaluate impact of impregnating mesh in .5% bupivacaine solution as compared to saline solution on length of hospital stay after laparoscopic ventral hernia repair.

Study Question:

Does impregnating mesh in solution of .5% bupivacaine before application in laparoscopic ventral hernia repair result in significant reduction in post-operative pain?

Null Hypothesis:

Post-operative pain after Impregnating the mesh before application in laparoscopic ventral hernia repair with 20 ml of 0.5% bupivacaine solution is either the same or more as compared to the post-operative pain after impregnating the mesh with 20ml of 0.9% saline solution.

Alternate Hypothesis:

Post-operative pain after Impregnating the mesh before application in laparoscopic ventral hernia repair with 20ml of 0.5% bupivacaine solution is less as compared to the post-operative pain after impregnating the mesh with 20ml of 0.9% saline solution.

Population:

Target Population:

Patients with un-complicated ventral abdominal wall hernia planned to undergo laparoscopic repair.

Study Population:

Patients with uncomplicated ventral abdominal wall hernia presenting at general surgery clinics of Aga Khan University Hospital (AKUH) Karachi and planned to have laparoscopic hernia repair.

Study Sample:

Patients with uncomplicated ventral abdominal wall hernia presenting at general surgery clinics of AKUH Karachi who are planned to undergo laparoscopic repair and meet eligibility criteria of inclusion into trial.

Randomization Technique:

Block randomization will be done. Blocks sizes each of 10 participants will be made. In each block randomization will be done using computer generated random numbers. Allocations in each block will be written on cards and enclosed in envelops. For each block envelops will be shuffled and then numbered in sequence. All envelops will be prepared and sealed before start of trial by clinical trial unit. Trial monitoring will be done by clinical trial unit. Emergency breaking of code will be done to the physician in cases of demanded for treatment of the patient.

SAMPLE SIZE:

Sample size was calculated using World Health Organization (WHO) software for sample size calculation. Muyosoms F et al in 2013 reported pain after laparoscopic ventral hernia repair after various mesh fixation techniques on visual analogue scale ranging from 0-10 . They reported pain after fixation with tackers to be 4.4 +/- 2.3 at four hours. It is hypothesized that bupivacaine soakage of mesh will reduce this pain by at least on third as compared to soakage with saline. A minimum of 44 patients are required in each group keeping level of significance of 5% and power of study to be 90%. Anticipating 10% loss to follow up, it was planned to include 50 patients in each group.

SETTINGS:

Study will be conducted in General Surgery Section of Aga Khan University Hospital, Karachi.

Patients will be evaluated in clinic at the time of presentation regarding eligibility to participate in study. Written informed consent will be taken in clinic. A copy of the consent form will be handed over to the patient. Clinical Trial Unit will be informed of the scheduled date and time of the operation. Allocation will be done by the staff at clinical trial unit which will be kept undisclosed to the investigators, patients and outcome assessors. Clinical Trial Unit will provide the solution for soaking mesh in coded form according to treatment arm allocation. After the operation first assessment of pain will be done six hours post-operatively using VAS. Second assessment will be done at twenty four hours from end of operation. This assessment will be done directly if patient is admitted in the hospital or will be done on telephone if patient is discharged home.

RECRUITMENT DURATION:

It is expected to complete recruitment of required sample size in one and a half year after start of trial.

Operative Procedure:

Laparoscopic ventral hernia repair is performed under general anesthesia. Laparoscopic approach to repair ventral hernia at our institution involves trans-abdominal approach through three laparoscopic ports inserted on one side of abdomen. Dual mesh is applied to anterior abdominal wall after reducing hernia contents. Mesh is soaked in saline before insertion into peritoneal cavity to ease handling. Mesh is applied using metallic tacks.

Trial Monitoring:

Bupivacaine is long acting local anesthetic drug. Though minimum toxic dose of bupivacaine for intra-peritoneal use is not defined, analgesic effect of its intra-peritoneal use especially after laparoscopic cholecystectomy has been assessed in several interventional studies. Intra-peritoneal use of up to 50ml of .25% , , or up to 20ml of .5% solution has not shown any drug related adverse reactions .

Known serious adverse reactions of bupivacaine after use as local anesthetic are due to its high serum concentrations after use, commonly seen after accidental administration directly into blood vessels. These are reported to be effects on central nervous system like seizures and convulsion and cardiac effects like arrhythmias and heart block. These adverse reactions are noted in 1:1000 cases . Time to onset of these adverse effects ranges from a few seconds to up to one hour . These adverse effects will be monitored for up to one hour after surgery in operating room and recovery room. In case some adverse effect is encountered, management will be done according to standard resuscitation protocols at our institution. Any adverse effect will be reported to Ethical Review Committee earliest after encountering and maximum of seven days after the event.

FOLLOW UP:

Pain assessment will be done using visual analogue scale (VAS). This is validated score to measure level of pain. It ranges from zero to ten. Score of 0 means no pain and score of ten means worst pain one can ever have. Score will be assessed at 6 and 24 hours from procedure.

ANALYSIS PLAN:

Intention to treat analysis will be done. Quantitative variable including VAS score will be reported in mean +/- standard deviation or median +/- interquartile range. Qualitative variables will be reported as percentages. Univariable linear regression will be done to assess linear association of VAS score with predictor variables including use of bupivacaine. Multiple variable linear regression analysis will be done to evaluate true effect of intervention, adjusting for time of assessment and amount of analgesia used. P value of less than 0.2 will be considered at Univariate level for the predictor variable to be included in multiple variable linear regression analysis. Possible effect modifiers like pre-operative pain and amount of dissection will be analyzed and reported if present.

Interim Analysis:

One interim analysis will be conducted in mid of trial. At the time of interim analysis, criteria to stop trial is defined as p value of less than 0.025 for the outcome of interest or less than .05 for adverse events like side effect of bupivacaine with power of 80%.

Linear Regression analysis will be done to adjust for confounders and effect modifiers.

Data Management:

Data will be collected on preformed printed questionnaires. Each questionnaire will be having information about data of operation and medical record number as identifier. Questionnaires will be anonymized and no identifiable information will be stored. Hard copies will be kept under lock and key in research office of Department of Surgery. Data will be entered in statistical software SPSS version 19. SPSS files will be password protected. Data will be stored till 15 year after completion of study.

ETHICAL CONSIDERATIONS:

Approval has been taken from Ethical Review Committee. Informed consent will be taken from participants. Cost of bupivacaine will be provided from study fund.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of age > 16 Years
* Both males and females
* Ventral Abdominal Wall Hernial Defect planned to undergo laparoscopic repair.
* Ventral Abdominal Wall Hernia is defined as defect in anterior abdominal wall through which contents of abdominal cavity can protrude. Anterior abdominal wall extends from Xiphisternum above to symphysis pubis below and anterior axillary lines laterally.
* We plan to include both primary and incisional hernias in our study.

Exclusion Criteria:

* Complicated Ventral Abdominal Wall Hernia (Strangulated, Obstructed)
* Recurrent Hernias
* Renal Insufficiency: Serum Creatinine > 1.5
* Hepatic Insufficiency: Known case of chronic liver disease or Total Bilirubin > 2mg/dl
* Pregnant or lactating Females
* Emergency Operations
* Current or regular use of analgesics for some other indication
* Patients with known hypersensitivity to the study drug.
* Refusal to Informed Consent
* Simultaneous additional surgical procedures

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-11-15 (Actual); Primary Completion 2017-04-30 (Estimated); Study Completion 2017-05-30 (Estimated)

PRIMARY OUTCOMES:
Post-Operative Pain will be graded on visual analogue scale (VAS) | Scale will be presented to the participant at 6 hours post procedure.
  Post-operative pain will be assessed by trained staff. Pain will be graded on visual analogue scale (VAS). VAS is validated scoring system according to which intensity of pain is scored on a scale of 0 to 10, 0 being no pain and 10 being worst pain.
Post-Operative Pain | Scale will be presented to the participant at 24 hours post procedure.
  Post-operative pain will be assessed by trained staff. Pain will be graded on visual analogue scale (VAS). VAS is validated scoring system according to which intensity of pain is scored on a scale of 0 to 10, 0 being no pain and 10 being worst pain.

SECONDARY OUTCOMES:
Length of hospital stay | Upto a maximum of 30 days from procedure
  Length of hospital stay will be taken in number of hours from time of end of operation till discharge from hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Tabish U Chawla, FRCS, Principal Investigator — Aga Khan University Hospital Karachi
Locations (1):
- Aga Khan University Hospital Karachi, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chawla T, Shahzad N, Ahmad K, Ali JF. Post-operative pain after laparoscopic ventral hernia repair, the impact of mesh soakage with bupivacaine solution versus normal saline solution: A randomised controlled trial (HAPPIEST Trial). J Minim Access Surg. 2020 Oct-Dec;16(4):328-334. doi: 10.4103/jmas.JMAS_50_19. PMID 32978352